CLINICAL TRIAL: NCT06298396
Title: A Prospective, Single Centre, Single-blinded, Within-subject Investigation, on the Effect of Stimulation Parameter Changes, and Monopolar and Dual-electrode Mode Changes, on Speech Perception in Experienced Adult Cochlear Implant Recipients
Brief Title: Investigating Stimulation Parameter and Electrode Mode Changes on Speech Perception in Experienced Adult Cochlear Implant Recipients
Acronym: DUAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5853
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Cochlear implant; Sensorineural hearing loss; Programming; Speech perception
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Masking Description: There is no masking in this study as all participants receive all MAPs (single group study model). The term "single-blinded" in the official title refers to the fact that participants are blinded to the order in which they receive the MAPs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAPs on Cochlear™ Nucleus® 7, Nucleus® 8 and Kanso® 2 Sound Processors (Experimental): Participants will receive four different MAPs to use during two take-home periods and will then complete hearing assessments using each MAP.
  Interventions: Device: Program using default MAP; Device: Program using low-power 1 (LP1) MAP; Device: Program using low-power 2 (LP2) MAP; Device: Program using low-power 3 (LP3) MAP

INTERVENTIONS:
Device: Program using default MAP — Each MAP uses a specific combination of stimulation parameters and electrode mode.
Device: Program using low-power 1 (LP1) MAP — Each MAP uses a specific combination of stimulation parameters and electrode mode.
Device: Program using low-power 2 (LP2) MAP — Each MAP uses a specific combination of stimulation parameters and electrode mode.
Device: Program using low-power 3 (LP3) MAP — Each MAP uses a specific combination of stimulation parameters and electrode mode.

SUMMARY:
This study aims to investigate the effect of stimulation parameters and different electrode modes on speech perception in adult cochlear implant recipients.

DETAILED DESCRIPTION:
Performance of four programs (MAPs), each with a different rate, PW and stimulation mode were evaluated, all using 8 maxima: (i) 900 Hz rate, 25 µs PW Default (ii) 900 Hz rate, 50 µs PW LP1, (iii) 500 Hz rate, 100 µs PW LP2 all using Monopolar stimulation mode, and (iv) 500 Hz rate, 100 µs PW using an investigational stimulation mode LP3

ELIGIBILITY:
Inclusion Criteria:

* Implanted with the CI600 Series (CI612, CI632, CI622, CI624), CI500 Series (CI512, CI513, CI532, CI522) or Freedom Series (CI24RE(CA), CI24RE(ST), CI24RE(CS), CI422)
* At least three months after activation of the cochlear implant.
* Eighteen years or older at the time of consent.
* User of 900Hz ACE (Advanced Combination Encoder) strategy MAP.
* Score of 20% or more for CNC words presented at 60dBSPL with CI alone in the test ear.
* Fluent speaker in English.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* One or more electrodes turned off in the MAP used regularly.
* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Current participation, or participation in another interventional clinical study/trial in the past 30 days, involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esti Nel, Principal Investigator — Cochlear
Locations (1):
- Cochlear Macquarie, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
Cochlear do not have an approved platform for public sharing of IPD collected in this study. Data may be provided to individual researchers on request.

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants evaluated each test of the 4 test programs:
  1. Default, 900 Hz stimulation rate (rate), 25 µs Pulse Width (PW) using Monopolar (MP) stimulation mode
  2. LP1, 900 Hz rate, 50 µs PW, MP mode
  3. LP2, 500 Hz rate,100 µs PW, MP mode
  4. LP3, 500 Hz rate, 100 µs PW, using an investigational stimulation mode
Period: Default MAP
Arm/Group | All Participants
Started | 20
Completed | 19
Not Completed | 1
Not completed — Protocol Violation | 1
Period: Low Power 1 (LP1) MAP
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0
Period: Low Power 2 (LP2) MAP
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0
Period: Low Power 3 (LP3) MAP
Arm/Group | All Participants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants were assigned to be tested with each test MAP (LP1, LP2, LP3) and the baseline (Default).
Groups:
- All Participants: All participants used four different MAPs (Default, LP1, LP2 and LP3) during two take-home periods, completing hearing assessments and questionnaires The study sound processor was Cochlear™ Nucleus® 7, Nucleus® 8 or Kanso® 2 sound processors depending on the participants usual Sound Processor type.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 15
Age, Continuous [Mean (Full Range); unit: years] | 70.2 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 20

OUTCOME MEASURES:

1. Primary Outcome: Paired Mean Difference Score for CNC Words Correct Between Default and LP1 MAPs in Quiet
Description: Speech perception in quiet was measured for each MAP using recorded CNC monosyllabic words.
  The goal of speech perception assessment in quiet was to compare % words correct for each of the conditions.
  The minimum score is 0% and maximum sore is 100%. A higher score means a better outcome.
  An average CNC word score for each MAP was calculated by combining the data from the specified timepoints.
Time Frame: 10 participants completed this test at Week 4, and 10 participants completed this at week 8
Population: One participant had the default MAP created using a Pulse Width of 37 µs rather than the required 25 µs, so there were 19 paired data points for analysis. All remaining participants were tested with the Default and LP1 MAPs
Measure: Mean (95% Confidence Interval); unit: percentage word score
Groups:
- Sound processor MAP: All participants were tested with each MAP
Arm/Group | Sound processor MAP
Number analyzed (Participants) | 19
percentage word score | -0.05 [-2.92 to 2.81]
Statistical Analysis 1: Comparison: Sound processor MAP; Test type: Non-Inferiority — A non-inferiority margin (NIM) of 10% was applied. In the sample size calculation, a 90% power to detect non-inferiority was used with a significance level α = 0.025 (one-tailed) was applied; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-2.92 to 2.81] — Treatment difference = LP1 - Default Non-inferiority demonstrated if the lower limit of the two-sided 95% confidence interval was above -10% (i.e. LP1 - Default > -10%)

2. Primary Outcome: Paired Mean Difference Score in dB SRT (AuSTIN) Between Default and LP1 MAPs in Noise
Description: Speech perception in noise was measured using the Australian Speech Test in Noise (AuSTIN), which is a test that uses recorded BKB-like target sentences.
  The goal of the speech perception test in noise is to provide the Speech Reception Threshold (SRT) in dB for 50% speech intelligibility (dB SRT) There is no minimum score. The maximum score is 15 dB. A lower score means a better outcome.
  An average SRT score for each MAP was calculated by combining the data from the specified timepoints.
Time Frame: 10 participants completed the test at Week 4, 10 participants completed the test at Week 8
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: dB SRT
Arm/Group | Sound processor MAP
Number analyzed (Participants) | 19
dB SRT | -0.32 [-0.87 to 0.24]
Statistical Analysis 1: Comparison: Sound processor MAP; Test type: Non-Inferiority — A non-inferiority margin (NIM) of 1 dB was applied. In the sample size calculation, a 90% power to detect non-inferiority was used with a significance level α = 0.025 (one-tailed) was applied; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.87 to 0.24] — The non-inferiority margin is 1 dB. Non-inferiority is demonstrated if the upper limit of the two-sided 95% confidence interval is < 1 dB

3. Secondary Outcome: Paired Mean Difference Score for CNC Words Correct Between LP1 and LP2 MAPs in Quiet
Description: Speech perception in quiet was measured for each MAP using recorded CNC monosyllabic words.
  The goal of speech perception assessment in quiet was to compare % words correct for each MAP.
  The minimum score is 0% and maximum sore is 100%. A higher score means a better outcome.
  An average CNC word score for each MAP was calculated by combining the data from the specified timepoints.
Time Frame: 10 participants completed the test at Week 4, 10 participants completed the test at Week 8
Population: All participants were tested with the LP1 and LP2 MAPs
Measure: Mean (95% Confidence Interval); unit: percentage word score
Arm/Group | Sound processor MAP
Number analyzed (Participants) | 20
percentage word score | 0.45 [-2.72 to 3.62]
Statistical Analysis 1: Comparison: Sound processor MAP; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.55 to 0.75] — Treatment difference = LP2 - LP1 Non-inferiority demonstrated if the lower limit of the two-sided 95% confidence interval was above -10% (i.e. LP2 - LP1 > -10%)

4. Secondary Outcome: Paired Mean Difference Score in dB SRT (AuSTIN) Between LP1 and LP2 MAPs in Noise
Description: as for outcome 2
Time Frame: 10 participants completed this test at Week 4, and 10 participants completed this at week 8
Population: All participants were tested with the LP1 and LP2 MAPs
Measure: Median (95% Confidence Interval); unit: dB SRT
Arm/Group | Sound processor MAP
Number analyzed (Participants) | 20
dB SRT | -0.23 [-0.55 to 0.75]
Statistical Analysis 1: Comparison: Sound processor MAP; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.55 to 0.75] — Treatment difference = LP2 - LP1 Non-inferiority demonstrated if the lower limit of the two-sided 95% confidence interval was < 1 dB (i.e. LP2- LP1 < 1 dB)

5. Secondary Outcome: Paired Mean Difference Score in Percentage CNC Words Correct Between LP1 and LP3 MAPs in Quiet
Description: as for outcome 1
Time Frame: 10 participants completed this test at Week 4, and 10 participants completed this at week 8
Population: All participants were tested with the LP1 and LP3 MAPs
Measure: Mean (95% Confidence Interval); unit: percentage word score
Arm/Group | Sound processor MAP
Number analyzed (Participants) | 20
percentage word score | -1.6 [-5.15 to 1.95]
Statistical Analysis 1: Comparison: Sound processor MAP; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.60, 95% CI 2-sided [-5.15 to 1.95]; Treatment difference = LP3 - LP1 Non-inferiority demonstrated if the lower limit of the two-sided 95% confidence interval was < 1 dB (i.e. LP3 - LP1 < 1 dB)

6. Secondary Outcome: Paired Mean Difference Score in dB SRT (AuSTIN) Between LP1 and LP3 MAPs in Noise
Description: as for outcome 2
Time Frame: 10 participants completed this test with at Week 4 and 10 participants completed this at week 8
Population: All participants were tested with the LP1 and LP3 MAPs.
Measure: Mean (95% Confidence Interval); unit: dB SRT
Groups:
- Sound processor: All participants were tested with each MAP
Arm/Group | Sound processor
Number analyzed (Participants) | 20
dB SRT | -0.39 [-1.10 to 0.32]
Statistical Analysis 1: Comparison: Sound processor; Test type: Non-Inferiority — non-inferiority margin (NIM) of 1 dB was applied. In the sample size calculation, a 90% power to detect non-inferiority was used with a significance level α = 0.025 (one-tailed) was applied; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.10 to 0.32] — Treatment difference = LP3 - LP1 Non-inferiority demonstrated if the lower limit of the two-sided 95% confidence interval was < 1 dB (i.e. LP3- LP1 < 1 dB)

7. Secondary Outcome: Switching Acceptability Rating Between LP2 and LP3 MAPs
Description: Participants rated the sound quality when switching between the LP2 and LP3 MAPs with the investigator asking the question: How does the sound quality of the new program compare with the previous program in terms of sound quality? The possible responses being "very different, somewhat different, similar, or the same". The number of participants in each category will be reported.
Time Frame: 10 participants were evaluated at week 4 and 10 participants were evaluated at week 8
Population: All participants evaluated switching between the LP2 and LP3 MAPs.
Measure: Count of Participants; unit: Participants
Arm/Group | Sound processor
Number analyzed (Participants) | 20
Participants
  Same sound quality | 5
  Similar sound quality | 8
  Somewhat different sound quality | 7
  Very different sound quality | 0

ADVERSE EVENTS:
Time Frame: Each participant was assessed from enrollment to final study visit, approximately 8 weeks
Groups:
- All Participants: All participants who were tested with each MAP and completed the study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=20)
Viral infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/96/NCT06298396/Prot_SAP_000.pdf